CLINICAL TRIAL: NCT02532907
Title: Study of Hepatic Responses in Patients Receiving Direct-acting Anti-HCV Drugs
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1794; UL1TR001082 (NIH)
Record Dates: First submitted 2015-08-13; First posted 2015-08-26 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Some of the data, blood and tissue that is taken during the study will be kept and used in future research to learn more about _Hepatitis C.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients who will have their second Liver biopsy at week 4: The 4 week time point is performed in lieu of the 12 week and the purpose of this time point is to evaluate earlier responses and transcriptional changes that might predict viral clearance or treatment failure in a subset of patients.
  Interventions: Procedure: Liver Biopsy
- Patients who will have their second Liver biopsy at week 12: Liver biopsies will be obtained at week 12 when most DAA treatments end in order to compare the hepatic responses induced or reduced by clearance of HCV
  Interventions: Procedure: Liver Biopsy

INTERVENTIONS:
Procedure: Liver Biopsy — patients will get a research liver biopsy pre-DAA treatment and either 4 or the standard 12 week time point. The liver biopsy is performed using standard protocol with ultrasound guidance.

SUMMARY:
This study is designed to obtain and store samples of serum and liver tissue in HCV (HepC Virus)-infected patients being treated with direct-acting antiviral (DAA) therapy, and to determine the effect of new DAA therapies on HCV-related responses in the liver and peripheral blood.

The introduction of new DAAs regimens that do not include IFN provides unique and novel opportunities to examine whether successful treatment-induced eradication of viral antigen results in reconstitution of T cell immunity. serum and liver tissue samples will be collected and stored in hopes of improving treatment and outcomes for future patients.

DETAILED DESCRIPTION:
This study is designed to obtain and store samples of serum and liver tissue in HCV-infected patients being treated with DAA therapy.

A liver biopsy will be performed pre-treatment for research reasons. A small liver sample that is not required for pathologic analysis will also be stored. Patients will undergo another liver biopsy at either 4 or 12 weeks after initiation of DAA therapy.

Any patients with HCV-related liver disease (age > 18) will be considered for this study.

Patients will have a 120 ml blood draw for research purposes at baseline and 12 weeks after stopping DAA treatment along with a 60 ml blood draw at 2, 4, 8, and 12 weeks of treatment.

The liver biopsy at baseline and then either at 4 or 12 weeks will be examined using molecular techniques to measure transcription of key genes involved in the antiviral response.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent
* Ages 18-70
* HCV-infected patients being treated with direct-acting antiviral (DAA) therapy.

Exclusion Criteria

* Pregnant women or females of childbearing potential that are not on contraception
* Institutionalized or mentally disabled persons
* Prisoners
* Unwilling or unable to provide informed consent
* Subjects who are HIV positive
* Anticipated inability to follow up
* Chronic anemia
* Platelet count < 100 for liver biopsy patients who have documented fatty liver disease by ultrasound prior to enrollment
* Any patient with bleeding disorders or prolonged INR
* Abstinent or consuming less than two drinks of alcohol per day.
* Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of patients will primarily occur through the Hepatology clinic, so non-veterans will be recruited. A total of 20 HCV-positive patients who will be treated with FDA-approved treatments as covered by the patient's insurance. Half of the patients will be treatment-naïve prior to enrollment and half will be treatment-experienced with either null response or relapse, i.e., persistent viremia. An equal proportion in each group will be biopsied at 4 versus 12 weeks after first dosing of DAA. Patients will be subjected to two biopsies during the life of the study.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Changes in gene array from baseline to either 4 or 12 weeks after treatment. | 1 year
  To examine the effect of new DAA therapies on HCV-related responses in the liver and peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Rosen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Sandra Boimbo, Aurora, Colorado, United States

REFERENCES:
- [Background] Golden-Mason L, Palmer B, Klarquist J, Mengshol JA, Castelblanco N, Rosen HR. Upregulation of PD-1 expression on circulating and intrahepatic hepatitis C virus-specific CD8+ T cells associated with reversible immune dysfunction. J Virol. 2007 Sep;81(17):9249-58. doi: 10.1128/JVI.00409-07. Epub 2007 Jun 13. PMID 17567698